CLINICAL TRIAL: NCT02056223
Title: Paracetamol Versus Ibuprofen for Patent Ductus Arteriosus Closure in Preterm Infants. A Prospective, Randomized, Controlled, Double Blind, Multicenter Clinical Trial.
Brief Title: Paracetamol vs Ibuprofen for PDA Closure in Preterm Infants.
Acronym: PARIDA
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: We enrolled only 53 patients
Sponsor: University of Padova (Other)
Responsible Party: Principal Investigator, Paola Lago, MD, University of Padova
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PARIDA 01/2013; 2013-004955-19 (EudraCT Number)
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Ductus Arteriosus Patent; Respiratory Distress Syndrome
Keywords: Patent ductus arteriosus; Preterm infant; Paracetamol; Ibuprofen
MeSH Terms: conditions — Ductus Arteriosus, Patent; Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- paracetamol (Experimental): Boluses of intravenous paracetamol at 15 mg/Kg four time a day for three consecutive days.
  Interventions: Drug: Intravenous paracetamol
- Intravenous ibuprofen (Active Comparator): Standard boluses of ibuprofen at 10-5-5-mg/Kg/dose once a day for three consecutive days.
  Interventions: Drug: Intravenous ibuprofen

INTERVENTIONS:
Drug: Intravenous paracetamol — 15 mg/Kg every 6 hours for three days
  Other Names: Paracetamol i.v.
  Arms: paracetamol
Drug: Intravenous ibuprofen — 10 -5-5 mg/Kg once a day for three days
  Other Names: Pedea i.v.
  Arms: Intravenous ibuprofen

SUMMARY:
Current pharmacological options to treat an hemodynamically significant PDA (HsPDA) in preterm infants are limited to non-selective cyclo-oxygenase (COX) inhibitors, indomethacin or ibuprofen. Recently paracetamol exposure has been reported to successful closure of PDA. Aim of this randomized double-blind controlled study is to compare the efficacy and the safety of standard PDA treatment ibuprofen versus paracetamol-experimental treatment . We hypothesize that paracetamol is more effective than ibuprofen in closing PDA, perhaps ameliorating the safety profile of the pharmacological treatment.

DETAILED DESCRIPTION:
The objective of this trial is to compare the efficacy and safety of 2 therapeutic regimens for PDA treatment in a population of preterm newborns of gestational age (GA) <31+6 weeks with respiratory distress syndrome (RDS) and HsPDA:

* Group A: experimental boluses of paracetamol at 15 mg/Kg four time a day for three consecutive days.
* Group B: standard boluses of ibuprofen at 10-5-5-mg/Kg/dose once a day for three consecutive days.

The primary objective of the study is: to evaluate the efficacy of paracetamol versus standard ibuprofen regimen, by comparing the rate of ductal closure after the first and second course of pharmacological treatment. (PDA diagnosed by ECHO criteria)

The secondary objective of the study is: to evaluate the safety of the above 2 therapeutic regimens in term of incidence of transient renal impairment, intraventricular hemorrhage (IVH) or other bleeding disorders, necrotizing enterocolitis (NEC) and isolated bowel perforation (without signs of NEC), incidence of sign of liver toxicity.

ELIGIBILITY:
Inclusion Criteria:

* inborn neonates
* preterm neonates ≤ 31+ 6 days weeks gestation
* newborns with HsPDA
* parental written informed consent for participation in the study must be obtained

Exclusion Criteria:

* Serum creatinine concentration greater than 1,5 mg/dl (132MMole/L)
* Urine output less than 1 ml/Kg/h
* Severe IVH (> grade II according to Volpe classification)
* Clinical bleeding tendency (as revealed by hematuria, blood in the gastric aspirate or in the stools, blood in the endotracheal tube aspirate)
* Necrotizing enterocolitis or marked abdominal distention with gastric bile residuals
* Thrombocyte count of less than 50.000/mm3
* Proved Sepsis
* Severe coagulopathy or liver failure
* Evidence of severe birth asphyxia, that is an APGAR score below 5 at 5 minutes of age and/or umbilical arterial pH < 7.0
* Known genetic or chromosomal disorders
* Participation in another clinical trial of any placebo, drug, biological, or device conducted under the provisions of a protocol.

Ages: 36 Hours to 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2017-01-09 (Actual); Primary Completion 2019-10-31 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
PDA pharmacological closure | Partecipants will be evaluated at the end of first and second course, at an expected avarage of 8 days of life (DOL)
  The rate of ductal closure after the first and second course of pharmacological treatment. (PDA diagnosed by ECHO criteria) in paracetamol versus ibuprofen group

SECONDARY OUTCOMES:
Oliguria | In the first 14 days of life
  Rate of oliguria defined as a reduction on urine output less than 1ml/Kg/h,

OTHER OUTCOMES:
Necrotizing enterocolitis (NEC) | In the first 14 days of life
  Rate of NEC in the paracetamol and ibuprofen group
Intraventricular haemorrhage (IVH) or death | Within 28 days of life
  Rate of intraventricular haemorrhage (IVH) or death within 28 days of life (composite outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Paola Lago, MD, Principal Investigator — Women's and Children's Health Department- AO- University of Padua
Locations (1):
- NICU, Women's and Children's Health Department, Azienda Ospedaliera-University of Padua, Padua, Italy

REFERENCES:
- [Result] Oncel MY, Yurttutan S, Degirmencioglu H, Uras N, Altug N, Erdeve O, Dilmen U. Intravenous paracetamol treatment in the management of patent ductus arteriosus in extremely low birth weight infants. Neonatology. 2013;103(3):166-9. doi: 10.1159/000345337. Epub 2012 Dec 19. PMID 23258386
- [Result] Hammerman C, Bin-Nun A, Markovitch E, Schimmel MS, Kaplan M, Fink D. Ductal closure with paracetamol: a surprising new approach to patent ductus arteriosus treatment. Pediatrics. 2011 Dec;128(6):e1618-21. doi: 10.1542/peds.2011-0359. Epub 2011 Nov 7. PMID 22065264
- [Result] Oncel MY, Yurttutan S, Uras N, Altug N, Ozdemir R, Ekmen S, Erdeve O, Dilmen U. An alternative drug (paracetamol) in the management of patent ductus arteriosus in ibuprofen-resistant or contraindicated preterm infants. Arch Dis Child Fetal Neonatal Ed. 2013 Jan;98(1):F94. doi: 10.1136/archdischild-2012-302044. Epub 2012 May 18. No abstract available. PMID 22611117
- [Result] Allegaert K, Palmer GM, Anderson BJ. The pharmacokinetics of intravenous paracetamol in neonates: size matters most. Arch Dis Child. 2011 Jun;96(6):575-80. doi: 10.1136/adc.2010.204552. Epub 2011 Feb 13. PMID 21317433